CLINICAL TRIAL: NCT03198221
Title: Randomized Comparison of the Impact of Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Versus Polyethylene Glycol Bowel Preparation on Inpatient Colonoscopy Quality Parameters
Brief Title: Comparison of Clenpiq vs Golytely Bowel Preparation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment due to difficult eligibility criteria and participant prep logistics
Sponsor: The Cleveland Clinic (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Carol Burke, MD, Staff, Department of Gastroenterology/Hepatology, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-127
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Bowel Preparation Solutions
Keywords: Golytely, Clenpiq, bowel prep
MeSH Terms: interventions — Golytely; polyethylene glycol 3350; Electrolytes; picosulfate sodium; Magnesium Oxide; Citric Acid

STUDY DESIGN:
Intervention Model Description: Participants will be receive either Golytely or Clenpiq bowel prep solutions. Both agents will either be administered as full dose the evening before or as split-dose on the evening before and on the day of the colonoscopy procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Active Comparator): Participants in Group A will begin drinking the bowel preparation Golytely (4 liter Polyethylene glycol based preparation) at 4:00 PM on the day before colonoscopy - an 8-ounce glass of the bowel preparation every 10 minutes. Participants must finish drinking the bowel preparation by 7:00 PM, and may continue to drink clear liquids until midnight.
  Interventions: Drug: Golytely
- Group B (Active Comparator): Participants in Group B will begin drinking the bowel preparation Golytely (4 liter Polyethylene glycol based preparation) at 4:00 PM on the day before colonoscopy - an 8-ounce glass of the bowel preparation every 10 minutes for a total of 8 glasses, and must complete drinking the bowel preparation by 5:30 PM. Participants may continue to drink clear liquids until midnight. The next day, 4 hours before the scheduled time of colonoscopy, participants will be asked to drink an 8 ounce glass of bowel preparation every ten minutes for a total of 8 glasses over no more than 1.5 hours. Participants may continue to drink clear liquids until 2 hours before the scheduled time of colonoscopy.
  Interventions: Drug: Golytely
- Group C (Active Comparator): Participants in Group C will begin drinking the bowel preparation Clenpiq (sodium picosulfate, magnesium oxide, and citric acid) at 4:00 PM on the day before colonoscopy. Participants will be asked to drink 5 ounces of the bowel preparation and at least five (5) additional 8-ounce glasses of clear liquids by 9:00 PM. At 10:00 PM, participants will drink another 5 ounces of the bowel preparation, and will then be asked to drink at least three (3) additional glasses of clear liquids by midnight.
  Interventions: Drug: Clenpiq
- Group D (Active Comparator): Participants in Group D will begin drinking the bowel preparation Clenpiq (sodium picosulfate, magnesium oxide, and citric acid) at 4:00 PM on the day before colonoscopy. Participants will be asked to drink 5 ounces of the bowel preparation and at least five (5) additional 8-ounce glasses of clear liquids by 9:00 PM, and may continue drinking clear liquids until midnight. The next day, 4 hours before the scheduled time of colonoscopy, participants will drink another 5 ounces of the bowel preparation and at least three (3) 8 ounce glasses of clear liquids within the next 2 hours. Participants may continue to drink clear liquids until 2 hours before the scheduled time of colonoscopy.
  Interventions: Drug: Clenpiq

INTERVENTIONS:
Drug: Golytely — bowel preparation
  Other Names: polyethylene glycol 3350 and electrolytes oral solution
  Arms: Group A; Group B
Drug: Clenpiq — bowel preparation
  Other Names: sodium picosulfate, magnesium oxide, anhydrous citric acid
  Arms: Group C; Group D

SUMMARY:
This is a prospective randomized study which will be done at main campus Cleveland Clinic. The investigators will be comparing the colon cleansing by the Boston Bowel Preparation Scale in participants undergoing colonoscopy as an inpatient at our hospital. Participants will be randomized to the the standard of care (4 Liter polyethylene glycol based preparation) or a low volume bowel preparation (sodium picosulfate, a stimulant laxative, magnesium oxide and anhydrous citric acid (SP/MC)). Both agents will either be administered as full dose the evening before or as split-dose on the evening before and on the day of the procedure.

DETAILED DESCRIPTION:
The purpose of our study is to determine if a 4L bowel cleansing agent is more effective than a low volume bowel preparation, and if the time of dosing (single dose night before vs split dose) of the bowel preparation results in better bowel cleansing in participants undergoing colonoscopy. Eligible participants undergoing colonoscopy with conscious sedation will be randomly assigned to one of two bowel preparations and one of two dosing schemas of bowel preparation. Participants not eligible for conscious sedation and are undergoing colonoscopy with general anesthesia will be randomized only to the single dose arms of the study. Participants will complete a questionnaire while drinking the bowel preparation to determine timing and tolerability of the bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

- Patients who need a colonoscopy while in the hospital (Cleveland Clinic main campus) will be eligible to participate.

Exclusion Criteria:

* Creatinine clearance less than 30 ml/min
* History of heart failure with current shortness of breath at rest causing limited physical activity, arrhythmia, unstable angina or acute myocardial infarction
* Small bowel obstruction, ileus or bowel perforation
* Dementia or cognitive dysfunction to an extent that they cannot perform the study related documentation or consent to participate in the study.
* Gastroparesis
* Toxic megacolon or undergoing colonoscopy for decompression
* Taking oral tetracyclines, fluoroquinolones, antibiotics, iron, digoxin, chlorpromazine and penicillamine within 2 hours before or 6 hours after administration of Clenpiq or stimulant laxatives within 24 hours
* History of prior colorectal surgery
* Allergy to any of the ingredients in Clenpiq or golytely
* if the procedure is planned in the intensive care unit (ICU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Burke, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 3 | 2 | 7 | 2
Completed | 3 | 2 | 7 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 3 | 2 | 7 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (12.7) | 42.5 (23.3) | 51.7 (21.9) | 58.0 (22.6) | 52.1 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 0 | 6
  Male | 1 | 1 | 4 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 3 | 2 | 6 | 1 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Satisfactory Bowel Cleansing
Description: Bowel cleansing efficacy will be measured using the Boston Bowel Prep Scale (BBPS). The BBPS divides the colon into 3 segments (right, transverse, left); each is scored from 0-3 (0=colonic mucosa not seen due to solid stool that cannot be cleared, 1=only a portion of the mucosa of the colon segment is seen due to staining, residual stool and/or opaque liquid, 2=minor amount of residual staining, small fragments of stool and/or opaque liquid but mucosa of colon segment is seen well, and 3=entire mucosa is seen well with no residual staining, small fragments of stool or opaque liquid). A total BBPS score of 6 or greater AND 2 or greater in all segments will be defined as satisfactory bowel prep. BBPS score of less than 6 or less than 2 in any segment of the colon will be taken as unsatisfactory bowel cleansing in the final analysis.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 3 | 2 | 7 | 2
Participants | 2 | 2 | 4 | 2

2. Secondary Outcome: Proportion of Participants Requiring a Repeat Colonoscopy
Description: Participants requiring a repeat procedure due to unsatisfactory bowel prep
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 3 | 2 | 7 | 2
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Data were collected over the space of 9 months
Description: Participants were observed for Adverse Events during the study procedure, and at any routine follow-up visits.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/7 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03198221/Prot_SAP_000.pdf